CLINICAL TRIAL: NCT04761614
Title: A Phase I Study of Riluzole in Combination With mFOLFOX6/Bevacizumab in Patients With Metastatic Colorectal Cancer
Brief Title: Riluzole in Combination With mFOLFOX6 and Bevacizumab in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ning Jin (Other)
Responsible Party: Sponsor-Investigator, Ning Jin, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-20096; NCI-2021-00018 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-01-21; First posted 2021-02-21 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Colorectal Carcinoma; Stage IV Colorectal Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Fluorouracil; dehydroftorafur; Leucovorin; Oxaliplatin; Riluzole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (riluzole, mFOLFOX6, bevacizumab) (Experimental): Patients receive riluzole PO BID on days 1-14. Patients also receive oxaliplatin via IVPB over 2 hours, leucovorin calcium IVPB over 2 hours, and bevacizumab IVPB over 30 minutes on day 1 and fluorouracil via IV push over 5 minutes and then IV continuously over 46 hours on days 1-2. Treatment repeats every 2 weeks for up to 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Fluorouracil; Drug: Leucovorin Calcium; Drug: Oxaliplatin; Drug: Riluzole

INTERVENTIONS:
Biological: Bevacizumab — Given IVPB
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-awwb; Bevacizumab-bvzr; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; Zirabev
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Leucovorin Calcium — Given IVPB
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Oxaliplatin — Given IVPB
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Drug: Riluzole — Given PO
  Other Names: Rilutek

SUMMARY:
This phase I trial is to find out the best dose, possible benefits, and/or side effects of riluzole and how well it works in combination with standard of care mFOLFOX6 and bevacizumab in treating patients with colorectal cancer that has spread to other places in the body (metastatic). Riluzole is a well-tolerated oral medication that has demonstrated it may make chemotherapy work better. Chemotherapy drugs, such as oxaliplatin, leucovorin calcium and fluorouracil, work in different ways to stop the growth of [cancer/tumor] cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Bevacizumab is an antibody that targets the blood vessel by blocking the activity of a protein called vascular endothelial growth factor alpha (VEGF-A). It helps to make the mFOLFOX6 more effective. Giving riluzole, mFOLFOX6, and bevacizumab may kill more tumor cells compared to mFOLFOX6 and bevacizumab alone in treating patients with colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Characterize the safety and toxicity of riluzole in combination with modified (m) leucovorin calcium, fluorouracil, and oxaliplatin (FOLFOX) 6/bevacizumab and determine the recommended phase II dose (RP2D) of riluzole in combination with mFOLFOX6/bevacizumab in patients with metastatic colorectal cancer.

SECONDARY OBJECTIVE:

I. Determine the pharmacokinetics of riluzole in patients with metastatic CRC.

EXPLORATORY OBJECTIVES:

I. Assess the efficacy of the combination treatment. II. Determine the effect of riluzole in downstream GRM3 signaling by immunofluorescent staining of phosphorylated (p)AKT and pCREB in pre- and post-treatment tumor tissues.

III. Assess FCGRT/FcRn expression, bevacizumab pharmacokinetics, inflammatory cytokines, and cachexia associated factors as early biomarkers for resistance to therapy.

IV. Assess cytotoxic T cells in peripheral blood to evaluate the immunomodulatory effect of this therapy.

OUTLINE: This is a dose-escalation study of riluzole.

Patients receive riluzole orally (PO) twice daily (BID) on days 1-14. Patients also receive oxaliplatin via intravenous piggyback (IVPB) over 2 hours, leucovorin calcium IVPB over 2 hours, and bevacizumab IVPB over 30 minutes on day 1 and fluorouracil via intravenous (IV) push over 5 minutes and then IV continuously over 46 hours on days 1-2. Treatment repeats every 2 weeks for up to 8 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic colorectal cancer, who are appropriate candidates to receive mFOLFOX6/bevacizumab. Patients who progressed on FOLFOX-based regimen are allowed
* Willingness to undergo both pre-treatment and post-treatment tumor tissue biopsies (pre-treatment tumor tissue will be sent to pathology lab to confirm metastatic colorectal cancer as the standard of care)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Age >= 18 years
* Absolute neutrophil count >= (ANC) 1,500/ul
* Platelets >= 100,000/ul
* Hemoglobin >= 9 g/dl
* Serum total bilirubin < 1.5 x ULN
* Serum albumin >= 2.5 g/dl
* If no liver involvement, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 1.5 x ULN. If liver involvement, AST and ALT =< 3.0 x ULN
* Ability to understand and the willingness to sign a written informed consent document
* A male subject of fathering potential must use an adequate method of contraception to avoid conception throughout the study (and for up to 12 weeks after the last dose of study drug) to minimize the risk of pregnancy. If the partner is pregnant or breastfeeding, the subject must use a condom
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 12 weeks after the last dose of study drug to minimize the risk of pregnancy. WOCBP must have a negative serum or urine pregnancy test within 72 hours before the start of the investigational product

Exclusion Criteria:

* Patients who are receiving any other investigational agents
* Patients with history of hepatitis B or C
* Patients with severe renal impairment (CrCl < 30 mL/min)
* Prior full field radiotherapy < 4 weeks or limited field radiotherapy < 2 weeks prior to first study drug administration. Patients with central nervous system (CNS) metastases may participate in this trial provided they are clinically stable. Patients who are < 1 month from radiation therapy must not be included
* Patients with existing grade 2 peripheral neuropathy
* Patients with a history of thrombotic or embolic events within the last six months such as a cerebrovascular accident (including transient ischemic attacks), pulmonary embolism or deep vein thrombosis
* Cardiac conditions as follows:

  * Active coronary artery disease, unstable or newly diagnosed angina or myocardial infarction less than 6 months prior to first study drug administration
  * Class III-IV New York Heart Association (NYHA) congestive heart failure
  * Uncontrolled hypertension (Systolic blood pressure [BP] > 150 mmHg and diastolic BP > 90 mmHg for 24 hours) despite optimal medical management
  * Corrected QT (QTc) (Friderica) prolongation > 480 msec
* Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, cardiac arrhythmia, active bleeding diatheses, and psychiatric illness/social situations that would limit compliance with study requirements
* Major surgical procedure or significant traumatic injury less than 3 weeks or those who receive minor surgical procedures within 1 week from first dose of study drug administration
* Known inability to swallow capsules
* Inability to comply with study and/or follow-up procedures
* Pregnant women are excluded from this study. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-05-06 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) | Up to 4 weeks (2 cycles of treatment) (1 cycle = 14 days)
  Will be defined by treatment related grade >= 4 adverse events or >= grade 3 alanine aminotransferase or aspartate aminotransferase elevation during the DLT period using the Common Terminology Criteria for Adverse Events version 5.0.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile of riluzole (Cmax) | Day 1 on cycle 1 (each cycle is 14 days)
  K data analysis will utilize a nonlinear mixed effects approach whereby PK parameter estimates will be generated from the data, and 'dose day' will be evaluated as a covariate on clearance and volume of distribution. The PK parameters including Cmax. Peak Plasma Concentration (Cmax)
Pharmacokinetic (PK) profile of riluzole (AUC) | Day 1 on cycle 1 (each cycle is 14 days)
  PK data analysis will utilize a nonlinear mixed effects approach whereby PK parameter estimates will be generated from the data, and 'dose day' will be evaluated as a covariate on clearance and volume of distribution. The PK parameters including AUC. Area under the plasma concentration versus time curve (AUC)

OTHER OUTCOMES:
Objective response rate (complete response + partial response) | Up to 112 days
  Will be estimated along with exact 95% confidence interval.
Change in phosphorylated (p)AKT and pCREB levels | Up to 42 days (each cycle is 14 days)
  Will be summarized using mean +/- standard error of mean, range, and median at each time point. Graphical analyses will be largely used to assess potential patterns and relationships.
Change in FCGRT/FcRn expression | Day 1 of cycle 1, 3, 5, 7 (each cycle is 14 days)
  Will be assessed using peripheral blood and summarized using mean +/- standard error of mean, range, and median at each time point. Graphical analyses will be largely used to assess potential patterns and relationships.
Change in bevacizumab clearance (Cmax) | Day 1 of cycle 1, 3, 5, 7 (each cycle is 14 days)
  Peak Plasma Concentration (Cmax)
Change in bevacizumab clearance (AUC) | Day 1 of cycle 1, 3, 5, 7 (each cycle is 14 days)
  Area under the plasma concentration versus time curve (AUC)
interleukin 6 | Day 1 of cycle 1 and day 1 of cycle 7 (each cycle is 14 days)
  Cytokines
leukemia inhibitory factor | Day 1 of cycle 1 and day 1 of cycle 7 (each cycle is 14 days)
  Cytokines
Necrosis factor alpha | Day 1 of cycle 1 and day 1 of cycle 7 (each cycle is 14 days)
  Cytokines
Interferon gamma | Day 1 of cycle 1 and day 1 of cycle 7 (each cycle is 14 days)
  Cytokines
C-reactive protein | Day 1 of cycle 1 and day 1 of cycle 7 (each cycle is 14 days)
  Cytokines
ferritin | Day 1 of cycle 1 and day 1 of cycle 7 (each cycle is 14 days)
  Cytokines
metalloproteinases 1 | Day 1 of cycle 1 and day 1 of cycle 7 (each cycle is 14 days)
  Cytokines
body weight | Day 1 of cycle 1 and day 1 of cycle 7 (each cycle is 14 days)
  Will include body weight and summarized using mean +/- standard error of mean, range, and median at each time point. Graphical analyses will be largely used to assess potential patterns and relationships.
skeletal muscle index | Day 1 of cycle 1 and day 1 of cycle 7 (each cycle is 14 days)
  Will include skeletal muscle index and summarized using mean +/- standard error of mean, range, and median at each time point. Graphical analyses will be largely used to assess potential patterns and relationships.
body serum albumin | Day 1 of cycle 1 and day 1 of cycle 7 (each cycle is 14 days)
  Will include body serum albumin and summarized using mean +/- standard error of mean, range, and median at each time point. Graphical analyses will be largely used to assess potential patterns and relationships.
Change in levels of circulating cytotoxic T cells | Day 1 of Cycle 1,3,5,7 (each cycle is 14 days)
  Will be assessed using peripheral blood mononuclear cells and summarized using mean +/- standard error of mean, range, and median at each time point. Graphical analyses will be largely used to assess potential patterns and relationships.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Jin, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT04761614/ICF_000.pdf